CLINICAL TRIAL: NCT05157997
Title: Transplantation of Deceased Donors With COVID-19 Into COVID-19 Negative Recipients Utilizing Casirivimab and Imdevimab Antibody Cocktail
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: New information regarding COVID-19
Sponsor: Northwell Health (Other)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 21-1223
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: COVID-19; Organ Transplant
Keywords: Regeneron; Covid-19 Antibodies
MeSH Terms: conditions — COVID-19 | interventions — casirivimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Casirivimab and Imdevimab Antibody Cocktail (Experimental): Patients receiving a Covid-19 positive liver, kidney, or heart transplant.
  Interventions: Drug: Casirivimab and Imdevimab Antibody Cocktail

INTERVENTIONS:
Drug: Casirivimab and Imdevimab Antibody Cocktail — The study will utilize REGEN-COV 8,000mg (4,000 mg of each monoclonal antibody) given as IV infusion on day of transplant and 2400mg (1,200 mg of each monoclonal antibody) on post-operative day 1.

SUMMARY:
This study will look to increase the donor pool for the solid organ transplant population by transplanting patients who died with COVID-19 but not from COVID-19 utilizing casirivimab and imdevimab antibody cocktail to prevent the transmission of the virus.

DETAILED DESCRIPTION:
This is single-center, proof of concept study that is expected to last up to three months. The target enrollment for this study is 14 subjects ≥18 years of age with a need of a kidney, liver or heart. This study will investigate the effects of the investigational product during a four-week intervention phase followed by a 12-month observation phase. Study population will be derived from patients in Northwell Health Transplant Center.

ELIGIBILITY:
Inclusion Criteria:

1. Subject provides written informed consent prior to initiation of any study procedures.
2. Understands and agrees to comply with planned study procedures.
3. Adult ≥18 years of age at time of enrollment, pediatric ages will be excluded.
4. Subject consents to receiving a COVID-19 positive organ (kidney, liver, or heart)

   a. Deceased immunocompetent donor with positive SARS-CoV-2 RT-PCR testing from the respiratory tract (upper or lower): i. Within 21 days since the date of COVID-19 diagnosis OR ii. Within 90 days since the date of COVID-19 diagnosis
5. Subject is confirmed COVID-19 negative confirmed by PCR at time of transplant with no signs and symptoms consistent with COVID-19
6. All candidates must be fully vaccinated 2 weeks prior to enrollment a. When applicable candidates can receive a booster vaccine as defined by the FDA/CDC

Exclusion Criteria:

1. Any exposure to investigational medications targeting COVID-19
2. Previous use of casirivimab with imdevimab antibody cocktail (REGEN-COV)
3. Previous treatment of COVID-19 with a monoclonal antibody
4. Active COVID-19 infection
5. Allergy to casirivimab with imdevimab
6. Pregnant patients
7. Prior transplant
8. Hepatitis C virus/NCT positive deceased donors

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Monitoring for SARS-CoV-2 infection | 30 days
  The overall objective of the study is to have transplant COVID-19 positive organs into COVID-19 negative recipients with no transmission of the virus. This will be assessed by monitoring for SARS-CoV-2 infection at different time points post-transplantation.

SECONDARY OUTCOMES:
30-day admission rate to hospital post-transplant due to COVID-19 | 30 days
  No 30-day readmission to the hospital due to COVID-19. All patients re-admitted to the hospital will be tested for COVID-19 by nasopharyngeal swab
Patient and graft survival at 30 days, 6 months and 1 year | 30 days, 6 months, and 1 year
  Assess patient and graft survival at 30 days
Adverse effects of casirivimab with imdevimab (REGEN-COV) antibody cocktail | 1 year
  Assessment of adverse effects of casirivimab with imdevimab
Stored serum will be evaluated when feasible for SARS-CoV-2 RNA | 30 days
  Biopsy proven rejection at 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Lewis Teperman, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Organ Transplant Center, Manhasset, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided